CLINICAL TRIAL: NCT05263024
Title: Study on the Significance of Auricular Clip in Prevention and Treatment of Valvular Heart Disease Atrial Thrombosis and the Related Precision Treatment Technique
Brief Title: Study on the Significance of Auricular Clip in Prevention and Treatment of Valvular Heart Disease Atrial Thrombosis
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-53-TYH
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Atrial Fibrillation; Thrombus; Embolism; Warfarin; Atrial Appendage; Surgery
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- left atrial appendage clip: Cardiac valvular patients complicated with atrial fibrillation need cardiac valvular surgery, according to the patient's wishes, cardiac auricular clamp at the same time
  Interventions: Device: atrial appendage clip
- Left atrial appendage treated with conventional methods: Valvular heart disease with atrial fibrillation requires valvular heart surgery and left atrial ligation
  Interventions: Device: atrial appendage clip

INTERVENTIONS:
Device: atrial appendage clip — During cardiac surgery, atrial fibrillation patients were treated with atrial appendage clipping

SUMMARY:
To evaluate the safety and clinical efficacy of left atrial appendage in the prevention of thrombus in patients with valvular heart disease, to improve the product according to clinical conditions, to achieve clinically accurate treatment, and to establish the heart valve, the usefulness and universality of Warfarin's anticoagulant model were verified by the specimen library

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common arrhythmia. The risk of ischemic stroke in AF patients is 4-5 times higher than that in non-af patients, and leads to nearly 20% mortality and nearly 60% disability. Atrial fibrillation is associated with valvular disease and atrial fibrillation in about 30-70% of patients with valvular heart disease. Left atrial thrombus occurs in 15-25% of patients with atrial fibrillation. More than 90% of patients with atrial thrombus is located in the left atrial appendage. In patients with valvular atrial fibrillation, the left atrial appendage is clamped at the same time of valvular surgery to avoid recurrence of atrial thrombus-related stroke. In this clinical trial, the left atrial appendage was used to clamp the prethrombotic site of the heart to prevent stroke and improve the prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with valvular heart disease aged between 18 and 75
2. Valvular heart disease [Cardiovascular Surgery Volume, Clinical Diagnosis and Treatment Guidelines, Chinese Medical Association (2011 edition)]
3. Preoperative cardiac function grade II-III (NYHA), no operation-related contraindications
4. Understand the nature of this study, agree to participate in all terms of this study, sign informed consent, agree to accept postoperative treatment plan and follow-up requirements, and cooperate to complete follow-up

Exclusion Criteria:

1. Patients whose left atrial appendage has been resected or occluded
2. She had a history of open heart surgery with extensive adhesion of the pericardium
3. Patients cannot be returned due to other reasons
4. Failed to reach the end point in clinical trials of other drugs or devices
5. X-ray is contraindicated or not suitable for TEE examination
6. Those who are considered unsuitable for the clinical trial by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients requiring heart valve surgery with atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2022-02-21 (Estimated); Primary Completion 2025-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Success rate of auricular clip clipping | 12 months
  Success rate of auricular clip clipping
Clinical success rate of auricular clip | 12 months
  Rate of patients without ischemic stroke, TIA, or systemic embolism 12 months after cardiac and auricular clipping

IPD SHARING:
Plan to Share IPD: No